CLINICAL TRIAL: NCT07380906
Title: Creation Of a Prospective Registry For Genicular Artery Embolization At The Joint & Vascular Institute
Brief Title: Prospective Registry For Genicular Artery Embolization At The Joint & Vascular Institute
Status: Recruiting | Type: Observational
Sponsor: Joint & Vascular Institute (Industry)
Responsible Party: Sponsor
Other Study IDs: 1396188
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthristis
Keywords: knee osteoarthritis; embolization; GAE; Genicular Artery Embolization
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Genicular Artery Embolization — Genicular Artery Embolization (GAE) is a minimally invasive, image-guided procedure in which embolic agents are delivered into hyperemic genicular arteries to reduce synovial inflammation and knee pain from osteoarthritis.

SUMMARY:
The goal of this observational study (prospective registry) is to collect long-term real-world data on the effectiveness and safety of genicular artery embolization (GAE) for knee osteoarthritis in adults aged 18 years or older with symptomatic KOA that has not responded to medical therapy.

The main questions it aims to answer are:

1. Does GAE lead to sustained improvement in pain (WOMAC, VAS) and quality-of-life scores over 12-36 months?
2. What patient or procedural factors are associated with better outcomes after GAE?

Participants will:

* Undergo GAE as part of their routine clinical care.
* Complete clinical follow-up assessments at 1, 3, 6, 12, 18, 24, and 36 months after treatment, including symptom and quality-of-life questionnaires.
* Have safety outcomes tracked according to Society of Interventional Radiology guidelines.

There is no comparison group; results will be analyzed to identify predictors of success and inform best practices for patient selection and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with symptomatic KOA refractory to medical therapy, referred for GAE.

Exclusion Criteria:

* Pregnancy, coagulopathy, severe comorbidities, or inability to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (18 years and older) presenting to the Joint & Vascular Institute for clinical consultation regarding symptomatic knee osteoarthritis. This population includes individuals who have failed standard medical management and are seeking minimally invasive alternatives to total knee arthroplasty. The registry will include men and women of all races and ethnicities without exclusion, provided they meet the clinical criteria for GAE as determined by the Principal Investigator or Sub-Investigators.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 5 years of enrollment/patient
  The investigators will describe differences in pain response with Genicular Artery Embolization (GAE) compared to a sham procedure when treating medically refractory mild to moderate Knee Osteoarthritis (KOA) at 12 months as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain subscale score. A higher score index a higher pain level while a lower score indicates lower pain levels. The score range is 0 to 96.

CONTACTS AND LOCATIONS:
Locations (1):
- Joint and Vascular Institute, Libertyville, Illinois, United States